CLINICAL TRIAL: NCT01543555
Title: Multicenter Randomized Controlled Trial of Loading Dose Statins for the Prevention of Cardiovascular Complications in High-Risk Non-Cardiac Surgery
Brief Title: Lowering the Risk of Operative Complications Using Atorvastatin Loading Dose
Acronym: LOAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Principal Investigator, Instituto de Ensino e Pesquisa, Research Institute HCor, Hospital do Coracao
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 02/15/2012
Record Dates: First submitted 2012-02-27; First posted 2012-03-05 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Myocardial Infarction; Peripheral Vascular Disease; Aortic Aneurism
Keywords: myocardial infarction; statin; perioperative care; peripheral vascular diseases; anesthesiology
MeSH Terms: conditions — Myocardial Infarction; Peripheral Vascular Diseases | interventions — Atorvastatin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin active (Experimental): Atorvastatin 80mg anytime within 18 hours before surgery. A postoperative 40mg atorvastatin dose administered at least 12 hours after the 80mg loading dose. Subsequently, 40mg atorvastatin daily for the next seven days.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Matching placebo 80mg anytime within 18 hours before surgery. A postoperative 40mg placebo dose administered at least 12 hours after the 80mg loading dose. Subsequently, 40mg placebo daily for the next seven days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80mg anytime within 18 hours before surgery. A postoperative 40mg atorvastatin dose administered at least 12 hours after the 80mg loading dose. Subsequently, 40mg atorvastatin daily for the next seven days.
  Other Names: Liptor (R); Kolevas (R)
  Arms: Atorvastatin active
Drug: Placebo — Matching placebo 80mg anytime within 18 hours before surgery. A postoperative 40mg matching placebo dose administered at least 12 hours after the 80mg loading dose. Subsequently, 40mg placebo daily for the next seven days.
  Other Names: Standard care
  Arms: Placebo

SUMMARY:
Patients submitted to noncardiac surgeries are at increased risk of serious cardiovascular complications. Statins have shown to lower cholesterol levels and reduce cardiovascular events in other scenarios. The objective of this study is to explore the effects of atorvastatin, as compared with placebo, on the 30-day risk of a composite of death, nonfatal Myocardial Injury after Noncardiac Surgery (MINS), or stroke among patients who undergo noncardiac surgery.

DETAILED DESCRIPTION:
Cardiovascular complications, such as myocardial infarction (MI) and stroke are common in the perioperative period of noncardiac surgeries. To the moment there are no safe and effective interventions to reduce vascular events in this scenario. Data from observational studies and small-sized randomized controlled trials (RCTs) have shown promising results in terms of risk reduction. In addition, experimental data have indicated that statins have acute anti-inflammatory properties, which promote the stabilization of atherosclerotic lesions and, therefore, might reduce the risk of MI, even in the short term. This study was designed to explore the effects of atorvastatin, as compared with placebo, on the 30-day risk of a composite of death, nonfatal Myocardial Injury after Noncardiac Surgery (MINS), or stroke among patients who undergo noncardiac surgery.

The study was conducted in accordance with the prespecified protocol and reached successful enrollment rates when, by the end of 2014 the steering committee was invited to join an international initiative and participate in a much larger clinical trial to investigate this relevant question. Due to this outstanding possibility, the steering committee decided to redesign the study which is now formatted as an exploratory trial. As described, the study was completed with the inclusion of 648 participants in June, 2015.

ELIGIBILITY:
Inclusion Criteria:

Patients older than 40 years-old undergoing non-cardiac surgery with an expected hospital stay of at least 24hs and that fulfills any one of the following criteria:

A) Established vascular disease:

i) Major vascular surgery ii) All types of surgery in patients with overt atherosclerosis (any significant or symptomatic coronary, cerebral or peripheral artery disease)

B) Without established vascular disease:

At least 3 risk factors for cardiovascular complications:

1. Major surgery;
2. Emergency surgery;
3. Previous history of heart failure;
4. diabetes;
5. Arterial hypertension;
6. Smoking habit along the last two years;
7. chronic kidney disease (creatinine greater than 2mg/dl);
8. Patients older than 70 years.

Exclusion Criteria:

* Previous intolerance to statins
* Current rhabdomyolysis
* Current use of statins
* Severe Liver Failure (CHILD-PUGH SCORE C)
* Breast-feeding or pregnancy
* Low-risk surgeries

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Composite outcome | 30 days
  Composite of all-cause mortality, nonfatal myocardial injury after noncardiac surgery and stroke at 30 days.

SECONDARY OUTCOMES:
All-cause mortality | 30 days
  Death from any cause.
Myocardial injury after noncardiac surgery (MINS) | 30 days
  An elevated cardiac troponin measurement judged due to cardiac ischemia (i.e., there was no evidence of a non-ischemic etiology like sepsis or pulmonary embolism).
Stroke | 30 days
  New neurologic symptom with compatible lesion on brain imaging and confirmation by a neurologist of the diagnosis of stroke.
Myocardial infarction | 30 days
  Rate of myocardial infarction as defined by any 2 of: typical chest pain OR typical ECG changes (ST-segment depression, ST-segment elevation, new Q waves, transitory T wave inversion) OR new rise in troponin levels (CK-MB levels if unavailable) OR new wall motion abnormality on echocardiogram. Pathological confirmation of myocardial necrosis on necropsy will also be accepted
Cardiovascular death | 30 days
  Evidence of death primarily caused by one of the following: acute myocardial infarction, stroke, pulmonary embolism, heart failure or ventricular arrhythmias.
Pulmonary embolism | 30 days
  Clinical signs accompanied by high-probability ventilation-perfusion lung scan or a filling defect of the pulmonary artery or its branches in a conventional arteriography or multi-slice spiral tomography.
Deep venous thrombosis | 30 days
  Any signs or symptoms of deep vein thrombosis confirmed by adequate images on ultrasound, computed tomography or angiography
Clinically relevant atrial fibrillation | 30 days
  A newly diagnosed atrial fibrillation that results in angina, heart failure, hypotension, or that requires treatment with an anti-arrhythmic drug or electric cardioversion
Rhabdomyolysis | 30 days
  elevation of CPK levels higher than 5 times the normal upper limit and myalgia or any CPK elevation higher than 10 times the upper limit, regardless of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Otávio Berwanger, MD, PhD, Study Chair — Hospital do Coração; Renato D Lopes, MD Phd, Study Chair — Brazilian Clinical Research Institute
Locations (1):
- Hospital do Coração, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] POISE Study Group; Devereaux PJ, Yang H, Yusuf S, Guyatt G, Leslie K, Villar JC, Xavier D, Chrolavicius S, Greenspan L, Pogue J, Pais P, Liu L, Xu S, Malaga G, Avezum A, Chan M, Montori VM, Jacka M, Choi P. Effects of extended-release metoprolol succinate in patients undergoing non-cardiac surgery (POISE trial): a randomised controlled trial. Lancet. 2008 May 31;371(9627):1839-47. doi: 10.1016/S0140-6736(08)60601-7. Epub 2008 May 12. PMID 18479744
- [Background] Kapoor AS, Kanji H, Buckingham J, Devereaux PJ, McAlister FA. Strength of evidence for perioperative use of statins to reduce cardiovascular risk: systematic review of controlled studies. BMJ. 2006 Dec 2;333(7579):1149. doi: 10.1136/bmj.39006.531146.BE. Epub 2006 Nov 6. PMID 17088313
- [Background] Durazzo AE, Machado FS, Ikeoka DT, De Bernoche C, Monachini MC, Puech-Leao P, Caramelli B. Reduction in cardiovascular events after vascular surgery with atorvastatin: a randomized trial. J Vasc Surg. 2004 May;39(5):967-75; discussion 975-6. doi: 10.1016/j.jvs.2004.01.004. PMID 15111846
- [Background] Dunkelgrun M, Boersma E, Schouten O, Koopman-van Gemert AW, van Poorten F, Bax JJ, Thomson IR, Poldermans D; Dutch Echocardiographic Cardiac Risk Evaluation Applying Stress Echocardiography Study Group. Bisoprolol and fluvastatin for the reduction of perioperative cardiac mortality and myocardial infarction in intermediate-risk patients undergoing noncardiovascular surgery: a randomized controlled trial (DECREASE-IV). Ann Surg. 2009 Jun;249(6):921-6. doi: 10.1097/SLA.0b013e3181a77d00. PMID 19474688
- [Background] Schouten O, Boersma E, Hoeks SE, Benner R, van Urk H, van Sambeek MR, Verhagen HJ, Khan NA, Dunkelgrun M, Bax JJ, Poldermans D; Dutch Echocardiographic Cardiac Risk Evaluation Applying Stress Echocardiography Study Group. Fluvastatin and perioperative events in patients undergoing vascular surgery. N Engl J Med. 2009 Sep 3;361(10):980-9. doi: 10.1056/NEJMoa0808207. PMID 19726772
- [Background] Patti G, Cannon CP, Murphy SA, Mega S, Pasceri V, Briguori C, Colombo A, Yun KH, Jeong MH, Kim JS, Choi D, Bozbas H, Kinoshita M, Fukuda K, Jia XW, Hara H, Cay S, Di Sciascio G. Clinical benefit of statin pretreatment in patients undergoing percutaneous coronary intervention: a collaborative patient-level meta-analysis of 13 randomized studies. Circulation. 2011 Apr 19;123(15):1622-32. doi: 10.1161/CIRCULATIONAHA.110.002451. Epub 2011 Apr 4. PMID 21464051